Official Title: Super-Supporters – Specially Trained Staff to facilitate Virtual Care for Vulnerable Patients and Family Caregivers: A real-world implementation and evaluation across North and South Carolina

NCT06841081

IRB Approved Date: 10/17/24



Department of Internal Medicine

# SUPER SUPPORTERS: SPECIALLY TRAINED STAFF TO FACILITATE VIRTUAL CARE FOR VULNERABLE PATIENTS AND FAMILY CAREGIVERS

Informed Consent Form to Participate in Research *Thomas Houston, MD,* Principal Investigators

## WHAT ARE THE RISKS OF THE STUDY?

The risk of harm or discomfort that may happen as a result of taking part in this research study is not expected to be more than in daily life or from routine physical or psychological examinations or tests. You should discuss the risk of being in this study with the study staff.

There is a slight risk of a breach of confidentiality. We will do our best to protect your confidential information. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe.

### ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

You are not expected to receive any direct benefit from taking part in this research study. We hope the information learned from this study will benefit other people in the future.

### WHAT ARE THE COSTS?

All study costs will be paid for by the study and costs for your regular medical care will be your own responsibility. As a thank you for your time, you will be paid \$20 for participating in the study.

#### WILL YOUR RESEARCH RECORDS BE CONFIDENTIAL?

The results of this research may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed unless it is authorized by you, required by law, or necessary to protect the safety of yourself or others. There is always some risk that even de-identified information might be re-identified.

## WHAT ABOUT MY PERSONAL INFORMATION?

In this research study, any new information we collect from you about your health or behaviors is considered <u>Protected Health Information</u>. The information we will collect for this research study includes: questions about your overall health and how you feel about interactions with your providers.

You can tell Dr. Thomas Houston that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:

#### **Thomas Houston**

Page 1 of 2
Adult Consent Form



However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.

WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

You may choose not to take part or you may leave the study at any time. Information about you may be removed from the study data and could be used for future research or shared with other researchers without additional consent from you.

If you have a question, you should contact the Chairman of the IRB at or the Research Subject Advocate at . You may also contact the Principal Investigator at .

By pressing continue, you agree to take part in this study. Participation is voluntary.

Page 2 of 2
Adult Consent Form